CLINICAL TRIAL: NCT02429518
Title: Dedicated QT Study in Bolivian Patients Taking Impavido® (Miltefosine) for Mucocutaneous Leishmaniasis
Status: Completed | Type: Observational
Sponsor: Knight Therapeutics (USA) Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MILT 2127-3
Record Dates: First submitted 2015-04-22; First posted 2015-04-29 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2019-03

CONDITIONS: Mucocutaneous Leishmaniasis
Keywords: leishmaniasis; miltefosine; EKG
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis | interventions — miltefosine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Miltefosine: Miltefosine: target of 2.5 mg/kg/day for 28 days
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine
  Other Names: Impavido

SUMMARY:
This study is a Phase 4, open-label, single group study in which at least 40 adult patients undergoing miltefosine treatment for mucocutaneous leishmaniasis (CL and ML) will be assessed by 12-lead ECG for prolongation of the corrected QT interval

DETAILED DESCRIPTION:
This study is a Phase 4, open-label, single group study in which at least 40 adult patients undergoing miltefosine treatment for mucocutaneous leishmaniasis will be assessed by digital 12-lead electrocardiogram (ECG) for prolongation of the corrected QT (QTc) interval. Potential subjects diagnosed with mucocutaneous leishmaniasis who are planning to undergo miltefosine treatment will be informed about the study and undergo the informed consent process. After obtaining informed consent, subjects will be screened over a 14-day period for eligibility by medical history including leishmaniasis diagnostics, physical examination, clinical laboratory measurements [chemistries: alanine aminotransferase (ALT), total bilirubin, creatinine, magnesium, calcium, potassium, sodium; hematology: white blood cell (WBC) count, hemoglobin, platelet count; and a pregnancy test if female], ECG, and medication use in the 28-day period before starting treatment. If eligible for the study, the subject will receive miltefosine for 28 days at a target dose of approximately 2.5 mg/kg/day. Screening and enrollment into the study will continue until at least 10 females and up to 30 males complete the study and are considered evaluable (provide Day 28 ECGs and pharmacokinetic (PK) samples and complete at least 25 of 28 days of miltefosine treatment). Vital signs will be collected weekly during treatment. Chemistries and hematology will be repeated at study Days 14 (mid-treatment) and 28 (end of treatment). A pregnancy test (if applicable) will be repeated at Day 28. ECGs (12-lead) will be repeated at Days 14 and 28. Blood will be drawn for PK assessments on Days 14 and 28 within 15 minutes of the final ECG. Adverse events (AEs) and concomitant medication use will be collected during treatment. If on Day 28, clinically significant abnormalities are observed by ECG, then a repeat ECG and PK blood draw will be performed at Day 42 (2 weeks after completing treatment). AEs and concomitant medication use will also be collected in any subject coming back for the Day 42 visit. Digital ECGs (12-lead) will be collected in triplicate at each time point over a period not to exceed 1 hour. During treatment, ECGs will be collected 4 hours after a dose (approximate Tmax).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Be available to complete study procedures
3. Have a diagnosis of mucocutaneous leishmaniasis confirmed by microscopy of a stained smear of a lesion sample, by culture of a lesion sample, or by polymerase chain reaction (PCR) of a lesion sample or by Montenegro skin test and be willing to undergo treatment with miltefosine
4. Be male or female and 18-55 years of age
5. Have alanine aminotransferase (ALT), total bilirubin, and creatinine < 1.5 x upper upper limit of normal (ULN)
6. Have white blood cell (WBC) count, hemoglobin, and platelet count within 15% of within normal limits (WNL)
7. Be without clinically significant non-cardiac medical disorder
8. Have 12-lead corrected QT interval using the Fridericia method (QTcF) interval < 450 msec, abnormal heart rate (< 40 or > 120 beats/min), PR interval (from 131 msec to 197 msec for males and 120 msec to 196 msec for females, or QRS interval (from 78 msec to 126 msec for males and 74 msec to 114 msec for females)
9. Have blood levels of ions that might affect ECG: (magnesium 1.82 mg/dL to 2.41 mg/dL, calcium 8.5 mg/dL to 10.5 mg/dL, potassium 3.5 milliequivalents/liter (mEq/L) to 10.5 mEq/L, and sodium 135 mEq/L to 148 mEq/L)
10. Have no family history of sudden cardiac death before age 40
11. Have no personal history ischemic heart disease, congestive heart failure, palpitations, dizziness, syncope, cardiac arrhythmias
12. If female, agree to use an effective method of birth control from the start of treatment until 5 months after completing treatment and have a negative pregnancy test

Exclusion Criteria:

1. Be a female who is breast feeding
2. Be a female who is pregnant
3. In the past 28 days prior to the start of miltefosine treatment have received any drug or other treatment that is known to significantly affect the QTc interval
4. Have positive serology for Chagas disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Persons with mucocutaneous leishmaniasis being treated with miltefosine
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
mean value of corrected QT interval | up to 2 weeks after end of treatment
  QTcF

SECONDARY OUTCOMES:
number of patients with adverse events | up to 2 months after end of treatment
  AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Soto, MD, Principal Investigator — Fundacion Nacional de Dermatologia
Locations (1):
- Funderma, Santa Cruz, Bolivia